CLINICAL TRIAL: NCT04923321
Title: Taste Supra-thresholds Among a Sample of Depressed Egyptian Adults Under Anti-depressants Therapy A Retrospective Cohort Study
Brief Title: Taste Supra-thresholds Among a Sample of Depressed Egyptian Adult Under Anti-depressants Therapy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christine Raouf George Mikhail, Principal Investigator, Cairo University
Other Study IDs: 18936
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Taste Disorders
MeSH Terms: conditions — Taste Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposure 1: commonly prescribed tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL) administered for at least 3 months
- Exposure 2: commonly prescribed Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine) administered for at least 3 months
- Non exposure: Non-pharmacological treatment (psychotherapy)

SUMMARY:
Determine the taste intensity at supra-threshold among a sample of depressed Egyptian adults (age from 20 to 50 years old) under anti-depressants therapy ( for at least 3 months) using filter paper disc(FPD) method using a psychophysical method through a scoring system.

DETAILED DESCRIPTION:
PECO

* P Population: depressed Egyptian adults under anti-depressants therapy
* E1 Exposure 1: Tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL)
* E2 Exposure 2: Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine)
* C control (non exposure) : non-pharmacological treatment ( psychotherapy)
* O Outcome: Determine the taste intensity at supra-threshold among these patients using a psychophysical method through a scoring system

ELIGIBILITY:
Inclusion Criteria:

* Depressed Egyptian adults under antidepressants therapy for at least 3 months/non-pharmacological treatment( psychotherapy) • Age from 20 to 50 years old

Exclusion Criteria:

* Antipsychotics

  * Hypnotics
  * Anticonvulsants
  * Ages other than the mentioned • Olfactory dysfunction
  * Chemosensory dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Depressed Egyptian adults under anti-depressants therapy The patients will be recalled using their phone numbers recorded in their follow up records in order to come to the Diagnosis center at the faculty of Dentistry, Cairo University to be assessed for taste intensity at supra-threshold level and will be given identification numbers and divided into three groups, to which the operator shall be blinded.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Taste intensity at supra-threshold | during a period of 3 months from February 2021 till April 2021]
  - C.M will assess the taste intensity at supra-threshold level on a 9 point vertical labeled scale (extremely strong, very strong, strong, slightly strong, neutral, slightly weak, weak , very weak, extremely weak) in which subjects indicate the intensity perceived when tasting a substance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No